CLINICAL TRIAL: NCT04606264
Title: Randomized, Embedded, Multifactorial Adaptive Platform for Perioperative Medicine at UPMC (UPMC REMAP): Core Protocol - Enhanced Recovery Protocols (ERP)
Brief Title: Recommendations of Enhanced Recovery Interventions for Patient's Clinical Team and Collection of Associated Data
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Holder-Murray (Other)
Collaborators: Berry Consultants (Other)
Responsible Party: Sponsor-Investigator, Jennifer Holder-Murray, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030022
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Perioperative Optimization
Keywords: perioperative; enhanced recovery; patient-directed care; randomized embedded multifactorial adaptive platform; REMAP; ERP; 90-day hospital free days; length of stay; perioperative optimization; oral morphine equivalents; postoperative nausea and vomiting; readmission
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Hydromorphone; Nerve Block; Perphenazine; Aprepitant; Dimenhydrinate; Ondansetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Major Abdominal: Neuraxial Analgesia (Active Comparator): Intrathecal morphine
  Interventions: Drug: Neuraxial Analgesia
- Major Abdominal: Regional Analgesia Block 1 (Active Comparator): Paravertebral block
  Interventions: Drug: Regional Block 1: Paravertebral
- Major Abdominal: PONV Optimal Prophylaxis (Active Comparator): Pre-op
  -perphenazine
  Induction -dexamethasone
  Emergence
  -ondansetron
  Interventions: Drug: Perphenazine; Drug: Ondansetron 4 MG; Drug: Dexamethasone
- Major Abdominal: PONV Supraoptimal Prophylaxis (Active Comparator): Pre-op
  * aprepitant
  * dimenhydrinate
  * perphenazine
  * ondansetron
  Induction -dexamethasone
  Emergence
  -ondansetron
  Interventions: Drug: Perphenazine; Drug: Aprepitant; Drug: Dimenhydrinate; Drug: Ondansetron 4 MG; Drug: Dexamethasone
- Major Abdominal: Regional Analgesia Block 2 (Active Comparator): QL1
  Interventions: Drug: Regional Block 2: QL1
- Major Abdominal: Neuraxial and Regional Analgesia Block 2 (Active Comparator): IT morphine and QL1
  Interventions: Drug: Neuraxial Analgesia; Drug: Regional Block 2: QL1
- Major Abdominal: Neuraxial and Regional Analgesia Block 1 (Active Comparator): IT morphine and paravertebral
  Interventions: Drug: Neuraxial Analgesia; Drug: Regional Block 1: Paravertebral

INTERVENTIONS:
Drug: Neuraxial Analgesia — This randomized group will receive a neuraxial morphine injection (intrathecal morphine/hydromorphone).
  Other Names: Intrathecal morphine/hydromorphone; IT morphine/hydromorphine
  Arms: Major Abdominal: Neuraxial Analgesia; Major Abdominal: Neuraxial and Regional Analgesia Block 1; Major Abdominal: Neuraxial and Regional Analgesia Block 2
Drug: Regional Block 1: Paravertebral — This randomized group will receive regional technique analgesia with sodium channel nerve blockade pharmacotherapy (ie nerve block)
  Other Names: Nerve Block
  Arms: Major Abdominal: Neuraxial and Regional Analgesia Block 1; Major Abdominal: Regional Analgesia Block 1
Drug: Perphenazine — This randomized group will receive 8 mg of perphenazine orally preoperatively.
  Arms: Major Abdominal: PONV Optimal Prophylaxis; Major Abdominal: PONV Supraoptimal Prophylaxis
Drug: Aprepitant — This randomized group will receive 40 mg of aprepitant orally preoperatively.
  Arms: Major Abdominal: PONV Supraoptimal Prophylaxis
Drug: Dimenhydrinate — This randomized group will receive 25 mg of dimenhydrinate orally preoperatively.
  Arms: Major Abdominal: PONV Supraoptimal Prophylaxis
Drug: Ondansetron 4 MG — This randomized group will receive 4 mg of ondansetron orally.
  Arms: Major Abdominal: PONV Optimal Prophylaxis; Major Abdominal: PONV Supraoptimal Prophylaxis
Drug: Dexamethasone — This randomized group will receive 4-5 mg of dexamethasone intravenously.
  Arms: Major Abdominal: PONV Optimal Prophylaxis; Major Abdominal: PONV Supraoptimal Prophylaxis
Drug: Regional Block 2: QL1 — This randomized group will receive regional technique analgesia with sodium channel nerve blockade pharmacotherapy (ie nerve block)
  Other Names: Nerve Block
  Arms: Major Abdominal: Neuraxial and Regional Analgesia Block 2; Major Abdominal: Regional Analgesia Block 2

SUMMARY:
This REMAP Periop ERP domain study falls under the Periop Core Protocol, which compares the different recommended strategies for enhancing recovery through the use of various standard of care treatments before, during and after surgery in all patients with elective surgical encounters at UPMC who meet eligibility criteria.

The ERP domain seeks to enhance recovery by optimizing strategies of perioperative care through evaluating combinations of perioperative treatment, which consists of preoperative, intraoperative and postoperative care. Optimal combinations of perioperative care will be generated and analyzed to determine the best outcomes for patients as defined by reduction in hospital free days, reduction in postoperative nausea and vomiting, and improved pain control.

DETAILED DESCRIPTION:
The Periop Core Protocol is an administration structure designed to provide appropriate management of all aspects of the study, taking into account multiple factors including representation from clinics and hospitals that are participating in the trial, availability of skills and expertise related to trial conduct and statistical analysis, and content knowledge regarding acute illness, elective surgery, and the interventions that are being evaluated. Eligible patients will be randomized to a recommended set of standard of care treatments related to their surgery to identify those that improve outcomes as defined by hospital free days at 30 days from the date of the surgical encounter. The administration model is designed to provide effective operational and strategic management of the REMAP that operates in multiple UPMC facilities, is supported by multiple funding bodies and sponsors, and will evolve with addition of domains and interventions that are being evaluated.

The ERP domain under the Periop Core Protocol will evaluate the varying recommended combinations of perioperative treatments, in hopes to determine the optimal strategies for perioperative care based on surgery type and patient specific factors. In this study, patient care components within the preoperative, perioperative, and postoperative domains will be randomized with a machine learning REMAP technique. Optimal strategies combining the entire perioperative process will be analyzed that determine best outcomes for patients including hospital free days, reductions in postoperative nausea and vomiting, and improved pain control.

ELIGIBILITY:
Inclusion Criteria

1. Patient is seen in preoperative appointment prior to surgery
2. ≥ 18 years of age
3. Anticipated overnight hospital stay
4. Scheduled for elective abdominal surgery that utilizes ERP PowerPlans - placed into the patient's electronic chart at least one night before surgery
5. ERP Abdominal Complex Pathway PowerPlan (used for colorectal and gastrointestinal surgery)
6. ERP Bariatric Surgery Pathway PowerPlan
7. ERP Gynecology Oncology Pathway PowerPlan
8. ERP Whipple/Pancreas Pathway PowerPlan
9. ERP Open Liver Resection Pathway PowerPlan
10. Surgery is scheduled for one of the following UPMC sites:
11. UPMC Presbyterian Hospital
12. UPMC Passavant Hospital
13. UPMC Magee-Women's Hospital

Exclusion Critera

1. Death is deemed to be imminent or inevitable
2. Patient is pregnant < 18 years of age
3. Patients undergoing emergent/urgent surgery
4. Patients that are pregnant
5. Patients that have an eligible PowerPlan ordered less than one night before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2977 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
30 day hospital free days | Day 0 - Day 30
  The primary endpoint for this domain is the REMAP Periop primary outcome of hospital free days at 30 days after the elective surgical encounter.

SECONDARY OUTCOMES:
Change in postoperative nausea and vomiting (PONV) by measurement incidences of emesis within 24 hours post surgery | 0 - 24 hours surgery
  Change in number of incidences of emesis 24 hours post surgery
Change in the rate of postoperative opioid use by measurement of oral morphine equivalents (OME) postoperative day 0 to postoperative day 1 | Day 0 - Day 1
  Change in the rate (mg/day) of Oral Morphine Equivalents administered

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Esper, MD, MBA, Study Chair — University of Pittsburgh
Locations (3):
- United States (3):
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data underlying the results reported in journal articles, subject to appropriate security controls, may be available for sharing with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Relevant data may be available 1 year following publication.
Access Criteria: Data access is subject to a methodically sound proposal and the necessary data sharing agreements.

REFERENCES:
- [Derived] Holder-Murray J, Esper SA, Althans AR, Knight J, Subramaniam K, Derenzo J, Ball R, Beaman S, Luke C, La Colla L, Schott N, Williams B, Lorenzi E, Berry LR, Viele K, Berry S, Masters M, Meister KA, Wilkinson T, Garrard W, Marroquin OC, Mahajan A. REMAP Periop: a randomised, embedded, multifactorial adaptive platform trial protocol for perioperative medicine to determine the optimal enhanced recovery pathway components in complex abdominal surgery patients within a US healthcare system. BMJ Open. 2023 Dec 28;13(12):e078711. doi: 10.1136/bmjopen-2023-078711. PMID 38154902